CLINICAL TRIAL: NCT06292533
Title: Effectiveness of Ultrapulse for the Treatment of Androgenic Alopecia Among Malaysian: A Quasi-experimental Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Yang Mooi Lim, Director (Institute of Postgraduate Studies and Research), Professor, Universiti Tunku Abdul Rahman
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTAR-30-2024
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Androgenic Alopecia; Alopecia
Keywords: Androgenic Alopecia; Alopecia treatment; Ultrapulse; Malaysian
MeSH Terms: conditions — Alopecia | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Ultrapulse treatment will be delivered by trained beautician for 6 sessions with 2 weeks interval. After the last session, participants will then follow up every 2 weeks for 1 month.
  Interventions: Device: Er:YAG laser
- Control-waitlist Group (No Intervention): Participants in control-waitlist group will receive homecare treatment that does not interfere with hair growth for 6 sessions with 2 weeks interval, follow up every 2 weeks for 1 month after last session and receive Ultrapulse treatment after the research end.

INTERVENTIONS:
Device: Er:YAG laser — Ultrapulse is a is a laser beauty device using erbium-doped yttrium aluminium garnet laser (er:YAG). Er:YAG laser is a laser with wavelength of 2940nm which is able to penetrate into the dermis to a depth of 3-4 mm, and energy absorption occurs in the area of the dermal papilla, resulting in an increase in blood circulation of the papilla and activation of metabolism in the hair follicle.
  Other Names: Ultrapulse
  Arms: Intervention Group

SUMMARY:
The goal of this study is to to evaluate the effectiveness of Ultrapulse for the treatment of androgenic alopecia among Malaysian. The main questions it aims to answer are:

* the efficacy of Ultrapulse in treatment of androgenic alopecia among Malaysian
* the safety and adverse effect of Ultrapulse treatment.
* the quality of life of androgenic alopecia among Malaysian.

DETAILED DESCRIPTION:
Ultrapulse is a is a laser beauty device using erbium-doped yttrium aluminium garnet laser (er:YAG). Er:YAG laser is a laser with wavelength of 2940nm which is able to penetrate into the dermis to a depth of 3-4 mm, and energy absorption occurs in the area of the dermal papilla, resulting in an increase in blood circulation of the papilla and activation of metabolism in the hair follicle. It generates multiple micro pores at the epidermal layer that enhances the absorption of the active substances that help to stimulate hair growth developed by Lyzer Co. Ltd in Korea.

ELIGIBILITY:
Inclusion Criteria:

- Patient with androgenic alopecia with severity of Norwood-Hamilton Scale II to VI for male and Ludwig Scale I to III for female

Exclusion Criteria:

* Use of topical or systemic medications affecting hair growth within the 6 months before recruitment
* Previous hair transplantation, underwent scalp reconstruction procedure, hair braiding or scalp tattoo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Global assessment of hair growth | 4 months
  Hair loss index will be recorded in the map and chart provided Cohen Hair Loss Classification System. The hair loss is scored with a single value from 1 to 100 to represent the percentage of hair of the patient's scalp.
  Global photography of the participant's scalp will be taken during first visit (baseline), immediate post-treatment (6 treatments), 2 weeks post-treatment and 1 month post-treatment.
  The evaluator will be responsible for scoring the hair loss index based on the global photograph provided.

SECONDARY OUTCOMES:
Patient satisfaction | 4 months
  The patient satisfaction of the participants in both intervention and control-waitlist group will be assessed during first visit (baseline), immediate post-treatment (6 treatments), 2 weeks post-treatment and 1 month post-treatment. by using SAPS questionnaire.
  It is scored by 0 (extremely dissatisfied) to 28 (extremely satisfied).
Quality of Life of Patient | 4 months
  The Hair specific Skindex-29 questionnaire comprised three types of scales: a symptom scale (7 items), a function scale (12 items), and an emotion scale (10 items). It is rated each question on a scale from 0 (never bothered) to 5 (always bothered). Responses for each item were converted to a linear scale, ranging from 0 (never bothered) to 100 (always bothered). A scale score represented the average score of the answered items, while a global score was the mean of the sums of each scale. A high score indicated a significantly impaired quality of life, whereas a low score indicated a mild impact on quality of life.
  The quality of life of the participants in both intervention and control-waitlist group will be assessed during first visit (baseline), immediate post-treatment (6 treatments), 2 weeks post-treatment and 1 month post-treatment.
Adverse effects | 4 months
  The adverse effects of the treatment will be recorded in the table in the provided sheet with the severity of 0 (no effect) to 3 (severe) except for pain using the visual analog scale from 0 (no pain) to 10 (extreme pain). The adverse effects will be recorded before and after participant received every treatment and during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Mooi Lim, PhD, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Hair Doc Puchong, Bandar Puchong Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dabek RJ, Austen WG Jr, Bojovic B. Laser-assisted Hair Regrowth: Fractional Laser Modalities for the Treatment of Androgenic Alopecia. Plast Reconstr Surg Glob Open. 2019 Apr 11;7(4):e2157. doi: 10.1097/GOX.0000000000002157. eCollection 2019 Apr. PMID 31321172
- [Background] Ke J, Guan H, Li S, Xu L, Zhang L, Yan Y. Erbium: YAG laser (2,940 nm) treatment stimulates hair growth through upregulating Wnt 10b and beta-catenin expression in C57BL/6 mice. Int J Clin Exp Med. 2015 Nov 15;8(11):20883-9. eCollection 2015. PMID 26885014
- [Background] Day D, McCarthy M, Talaber I. Non-ablative Er:YAG laser is an effective tool in the treatment arsenal of androgenetic alopecia. J Cosmet Dermatol. 2022 May;21(5):2056-2063. doi: 10.1111/jocd.14370. Epub 2021 Aug 26. PMID 34435735
- [Background] Han SH, Byun JW, Lee WS, Kang H, Kye YC, Kim KH, Kim DW, Kim MB, Kim SJ, Kim HO, Sim WY, Yoon TY, Huh CH, Hwang SS, Ro BI, Choi GS. Quality of life assessment in male patients with androgenetic alopecia: result of a prospective, multicenter study. Ann Dermatol. 2012 Aug;24(3):311-8. doi: 10.5021/ad.2012.24.3.311. Epub 2012 Jul 25. PMID 22879715